CLINICAL TRIAL: NCT02348671
Title: Evaluation of Wound Dressings to Reduce the Harmful Effects of Shear- Force at the Skin
Brief Title: Evaluation of Wound Dressings in the Reduction of Shear- Force
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SF-2
Record Dates: First submitted 2014-12-01; First posted 2015-01-28 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-01

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: shear- force — 19 Newton shear- force and 3,9 kPa pressure for half an hour

SUMMARY:
The purpose of this study is to investigate if wound dressings are capable in reducing the effects of shear- force at the skin. With our own shear- force model we are able to apply 19 Newton shear- force combined with 9 newton pressure at the skin of the non- dominant forearm. After half an hour we measure IL-1alpha/ total protein- ratio, cutaneous blood flow (Laser doppler, Moor LDI) and the erythema index (DSMIIColormeter) which occurs as an effect of shear- force application at the skin.

Then, we apply 19 Newton shear- force combined with 9 Newton pressure at the dominant fore-arm but this time we put a wound dressing between the skin and shear- force model. After half an hour we measure the IL-1alpha/total protein-ratio, cutaneous blood flow and the erythema index.

This research consists of three research day, each day we are going to investigate a different wound dressing

ELIGIBILITY:
Inclusion Criteria:

* healhty volunteer
* age 18- 30
* BMI 20- 30

Exclusion Criteria:

* Trauma fore-arms
* Diabetes mellitus type I or type II
* The use of NSAID's in the last 7 days
* Vascular diseases
* Muscular dystrophy
* Malignancy
* Participant is unable to give informed consent

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ten healthy volunteers
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Cutaneous blood flow, erythema index, IL-1alpha/Total protein ratio | Directly after intevention